CLINICAL TRIAL: NCT01291966
Title: Efficacy of a Intervention to Reduce Medication Errors and Therapeutic Failure in Patients Over 65 Years Polypharmacy
Brief Title: Efficacy of a Intervention to Reduce Medication Errors and Improve Adherence
Acronym: ATEM-AP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Collaborators: Sociedad Andaluza de Medicina Familiar y Comunitaria (Unknown); Sociedad Española de Medicina Familiar y Comunitaria (Unknown)
Responsible Party: Luis A Pérula, Andalusian Health Service
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI-0101/2008
Record Dates: First submitted 2011-01-26; First posted 2011-02-09 (Estimated); Last update posted 2011-02-09 (Estimated); Status verified 2010-12

CONDITIONS: Medication Adherence; Patient Compliance
Keywords: medication errors; Patient Compliance; patient safety; polypharmacy
MeSH Terms: conditions — Medication Adherence; Patient Compliance | interventions — Motivational Interviewing; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Motivational interview (Experimental)
  Interventions: Behavioral: Motivational interview

INTERVENTIONS:
Behavioral: Motivational interview
  Other Names: Counseling; Patient-centered method

SUMMARY:
The purpose of this study is to demonstrate that an intervention based on the motivational interview directed to patients with polypharmacy to improve the Therapeutic Adherence and to reduce the errors of Medication in major measure that the habitual intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with polypharmacy (5 or more medicines)
* That detects to them a problem of Therapeutic Adherence
* That agree to take part in the study

Exclusion Criteria:

* Immobilized patients or with an index of Barthel lower than 60 points
* Incapable to fulfill ABVD
* Patients with cognitive deterioration
* Patients with diagnosis of ictus in the last 6 months
* That has been admitted to hospital 2 or more times in the last year Institutionalized patients

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 154 (Actual)
Dates: Start 2010-01; Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
medication errors in the patients | Baseline, 1, 3 and 6 months
  Medication errors before and after the intervention in each group

SECONDARY OUTCOMES:
Percentage of adherence | Baseline and 6 months
  To measure adherence to treatment will use a combination of direct methods (counting of medication) and indirect tests are passed or self-reported compliance test Haynes-Sackett and Morisky-Green test

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Perula, PH D, Principal Investigator — Andalusian Health Service
Locations (1):
- Unidad Docente de Medicina Familiar y Comunitaria, Córdoba, Córdoba, Spain

REFERENCES:
- [Derived] Moral RR, Torres LA, Ortega LP, Larumbe MC, Villalobos AR, Garcia JA, Rejano JM; Collaborative Group ATEM-AP Study. Effectiveness of motivational interviewing to improve therapeutic adherence in patients over 65 years old with chronic diseases: A cluster randomized clinical trial in primary care. Patient Educ Couns. 2015 Aug;98(8):977-83. doi: 10.1016/j.pec.2015.03.008. Epub 2015 Mar 18. PMID 25858633
- [Derived] Perula de Torres LA, Pulido Ortega L, Perula de Torres C, Gonzalez Lama J, Olaya Caro I, Ruiz Moral R; Grupo corporativo Estudio ATEM-AP. [Efficacy of motivational interviewing for reducing medication errors in chronic patients over 65 years with polypharmacy: Results of a cluster randomized trial]. Med Clin (Barc). 2014 Oct 21;143(8):341-8. doi: 10.1016/j.medcli.2013.07.032. Epub 2013 Dec 28. Spanish. PMID 24378144